CLINICAL TRIAL: NCT05085899
Title: Physical Fitness Normative Values Among School Going Children
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Sana Manzoor
Record Dates: First submitted 2021-08-20; First posted 2021-10-20 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Physical Fitness; Cardiorespiratory Fitness
Keywords: Normative values; Cardiorespiratory Fitness; School Going Children

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Physical fitness is state of health and wellbeing, it determines ability of body to perform sports or daily physical activities. Physical fitness is related to our cardiorespiratory fitness level, as cardiorespiratory fitness levels used for decreasing chronic diseases, promoting overall cardiovascular and general body health, decreasing the chance of developing disorders due to poor physical fitness. Different tests will be used for the measurement of physical fitness in school going children such as 1. height and weight, 2.waist circumference, 3.triceps skinfold thickness, 4.subscapular skinfold thickness, 5.standing long jump test, 6.handgrip strength test, 7. 20 m shuttle run test, 8. 4x10 m shuttle run test.

This study will be Cross-sectional study and will be conducted in schools in order to determine physical fitness level in school going children and adolescents between age 10-17-year-old. Data will be collected by non-probability convenience sampling technique. Early determination of physical fitness level in school going children will be helpful, to promote their health status and to prevent the incidence of cardiovascular disorders.

DETAILED DESCRIPTION:
Evidence shows that low physical fitness level and cardiorespiratory level are strongly and independently associated with high risk of cardiovascular disorders, diabetes, mental health, stroke other risk factors and comorbidities. In children and adolescents, peak oxygen uptake (VO2peak) is the most researched physiological variable in pediatric exercise physiology for its association with cardio-metabolic risk factors and other health-related variables . Children's health and well-being is highly correlated with their physical fitness. Recently published studies indicate that low levels of physical fitness (e.g., cardiorespiratory fitness, muscular endurance/power) are associated with an elevated risk of developing adverse physiological events (e.g., unbalanced body mass index, waist circumference, systolic blood pressure, plasma glucose, lipoprotein cholesterol, insulin resistance) in school-aged students.

Physical fitness is usually determined in school-aged children using health-related physical fitness batteries (i.e., field tests). Compared to more sophisticated laboratory-based test equipment, field tests are easy-to-administer, involve minimal equipment and personnel, demonstrate good validity and reliability and a large number of subjects can be tested in a relatively small amount of time. Normative data derived from field tests have previously been used to identify subjects for health/talent promotion or to provide current objective recommendations for the assessment of physical fitness during physical education.

In this study investigator will determine physical fitness normative values in school going children, in order to determine present health status which will reduce the incidence of future occurrence of cardiovascular disorders. Present health status is strong predictor of future cardiovascular disorders.

ELIGIBILITY:
Inclusion Criteria:

School going children of age 10-18 years,

Exclusion Criteria:

* Mentally unstable children
* Children having any disorders

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Physical fitness will be measured by ALPHA health related fitness test battery in children and adults. Following tests will be used to determine normative values of physical fitness such as,
  1. Morphological components
  2. Waist circumference
  3. Subscapular skinfold
  4. Triceps skinfold.
  5. Musculoskeletal component
  6. Standing broad jump
  7. 4x10 m run test
  8. 20m shuttle test
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
ALPHA Health-Related Fitness Test Battery for Children and Adolescents | Day 1
  The ALPHA fitness test battery is a developed tool to provide a set of valid, reliable, feasible and safe field-based fitness tests for the assessment of health-related physical fitness in children and adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos-Sepulveda JA, Ramirez-Velez R, Correa-Bautista JE, Izquierdo M, Garcia-Hermoso A. Physical fitness and anthropometric normative values among Colombian-Indian schoolchildren. BMC Public Health. 2016 Sep 13;16(1):962. doi: 10.1186/s12889-016-3652-2. PMID 27619491
- [Background] Lesinski M, Schmelcher A, Herz M, Puta C, Gabriel H, Arampatzis A, Laube G, Busch D, Granacher U. Maturation-, age-, and sex-specific anthropometric and physical fitness percentiles of German elite young athletes. PLoS One. 2020 Aug 13;15(8):e0237423. doi: 10.1371/journal.pone.0237423. eCollection 2020. PMID 32790710
- [Background] Ramirez-Velez R, Silva-Moreno C, Correa-Bautista JE, Gonzalez-Ruiz K, Prieto-Benavides DH, Villa-Gonzalez E, Garcia-Hermoso A. Self-Rated Health Status and Cardiorespiratory Fitness in a Sample of Schoolchildren from Bogota, Colombia. The FUPRECOL Study. Int J Environ Res Public Health. 2017 Aug 23;14(9):952. doi: 10.3390/ijerph14090952. PMID 28832546
- [Background] Thomas E, Petrigna L, Tabacchi G, Teixeira E, Pajaujiene S, Sturm DJ, Sahin FN, Gomez-Lopez M, Pausic J, Paoli A, Alesi M, Bianco A. Percentile values of the standing broad jump in children and adolescents aged 6-18 years old. Eur J Transl Myol. 2020 Jun 17;30(2):9050. doi: 10.4081/ejtm.2019.9050. eCollection 2020 Jul 13. PMID 32782766
- [Background] Godoy-Cumillaf A, Bizzozero-Peroni B, Tomkinson GR, Brazo-Sayavera J. Physical fitness of Latin America children and adolescents: a protocol for a systematic review and meta-analysis. BMJ Open. 2021 May 3;11(5):e047122. doi: 10.1136/bmjopen-2020-047122. PMID 33941634